CLINICAL TRIAL: NCT04976374
Title: A Multimodal Analgesic Protocol With Gabapentin Dexmedetomidine For Postoperative Pain Managment After Modified Radical Mastectomy Surgery: A Randomized Placebo-Controlled Study
Brief Title: Analgesic Protocol With Gabapentin Dexmedetomidine For Postoperative Pain Managment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Ahmed Bakir, Assistant Professor of Anesthesia, Intensive care and Pain Relief, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AP2105-50105
Record Dates: First submitted 2021-07-05; First posted 2021-07-26 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexmedetomidine; Gabapentin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients of group A will start dexmedetomidine (precedex 100 ug lmL, Hospira) infusion 0.4 ug {Kg}h after bolus of 0.5 ug 1 kg intravenously over 10 min
  Interventions: Drug: Dexmedetomidine and Gabapentin
- Group B (Placebo Comparator): Group B will recive a bolus of saline then saline infusion identical to group A
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Dexmedetomidine and Gabapentin — Administration of intravenous dexmedetomedine for post operative analgesic purposes in combination with gabapentin
  Other Names: gabapentin
  Arms: Group A
Other: Saline — Intravenous Saline 0.9% for placebo purposes
  Arms: Group B

SUMMARY:
Assessment of quality of post mastectomy analgesic protocol of Gabapentin and Dexmedetomedine in a placebo-controlled study

DETAILED DESCRIPTION:
Assessment of quality of post mastectomy analgesic protocol of Gabapentin and Dexmedetomedine in a placebo-controlled study.

Dexmedetomidine is a highly selective X2 adrenergic receptor aganist; it has anxiolytic, sedative, analgesic and sympathdytic properties without significant respiratory depressant effects. Research evidence has shown that this drug protects the body (including heart, nerves, etc.) against ischemia and hypoxic injury. Therefore, dexmedetomidine can be one of the best options for reducing pain after surgery.

Gabapentin, a structural analog of gamma aminobutyric acid, is used as an anticonvulsant drug since 1993. In addition it has been effective in neuropathic pain, diabetic neuropathy and reflex sympathetic dystrophy. It acts through binding to the X-2-5 subvnits of voltagegated calcium ion channels and preventing the central sentization and hyperalgesia. Gabapentin has demonstrated to inhibit the development and establishment of hyperalgesia and secondry allodynia in human volunteers.

Gabapentin may also decrease postoperative obioid requirement through preventing the tolerance development. Furthermore, it has minimal or no effect on gastric mucosa, renal function, and platelets count or activity in the perioperative period to be prefer over nonsteroidal anti-inflammatory drugs.

The Combination of both drugs will be tested for potentiation of post-operative analgesia and decrease of opioid consumptions

ELIGIBILITY:
Inclusion Criteria:

* adult female patients below 65 years of age scheduled for modified radical mastectomy surgery, American society of Anesthesiologists(ASA) physical status I-II

Exclusion Criteria:

* known allergy to study drugs; patients already taking oral gabapentin, knal or hepatic defunction, current treatment with narcotics, antihypertensives, benzodiazepines, X2 agonists, antiepileptics and antipsychotics

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-11-25 (Estimated); Study Completion 2021-11-25 (Estimated)

PRIMARY OUTCOMES:
Post operative morphine consumption | 24 hours
  Evaluation of the effects of combining and gabapentin and dexmedetomidine infusion on post operative morphine consumption within the first 24 h in patients undergoing modified radical mastectomy surgery

SECONDARY OUTCOMES:
Post operative VAS score | 24 hours
  Evaluation of the effects of combining and gabapentin and dexmedtomidine infusion on post operative visual analogue scale (VAS) score within the first 24 h in patients undergoing modified radical mastectomy surgery

CONTACTS AND LOCATIONS:
Locations (1):
- NCI Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol, methodology and results to be shared with other researchers